CLINICAL TRIAL: NCT00814957
Title: An Open Label Positron Emission Tomography Study in Healthy Male Subjects to Investigate Brain Dopamine D3 Receptor Occupancy, Pharmacokinetics and Safety of Single Oral Doses of GSK618334, Using 11C-PHNO as PET Ligand.
Brief Title: An Open Label Positron Emission Tomography (PET) Study of GSK618334 in Healthy Male Subjects Using 11C-PHNO as PET Ligand
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110269
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Substance Dependence
Keywords: positron emission tomography; addiction
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label (Experimental): D3 receptor antagonist
  Interventions: Drug: GSK618334

INTERVENTIONS:
Drug: GSK618334 — D3 receptor antagonist

SUMMARY:
The purpose of this study is to investigate the relationship between the plasma concentrations of the study drug and the amount of the study drug bound to the D3 receptors of the brain after dosing of a new compound GSK618334.

DETAILED DESCRIPTION:
This imaging study will be an open label, non-randomised PET receptor occupancy study using healthy male volunteers. The time course and degree of D3 receptor occupancy (RO) after single doses of GSK618334 will be determined using 11C-PHNO as a PET ligand labeling dopamine receptor. The PK/PD relationship between plasma concentrations of GSK618334 and D3 RO will be described. Potential relationships between D3 RO and functional magnetic resonance imaging (fMRI) endpoints will be assessed as an exploratory aim.

ELIGIBILITY:
Inclusion Criteria:

* healthy, male subjects aged between 30 and 55 old inclusive.
* normal body weight.
* normal ECG and vital signs.
* agree to use acceptable contraceptive methods required.
* capable of giving written informed consent.

Exclusion Criteria:

* smoker or uses other nicotine-containing products.
* certain medical conditions including heart disease, neurological disease, gastrointestinal disease, kidney or liver dysfunction - abnormal laboratory tests.
* certain psychiatric conditions and use of certain psychoactive drugs .
* positive blood alcohol or urine drug test.
* alcohol intake over 14 drinks per week.
* participation in another drug trial within 30 days or a study involving significant radiation exposure.
* donation of more than 450 mL blood within the 56 days.
* family history of cancer (one or more first-degree relative diagnosed before the age of 55 years old).
* having cardiac pacemaker or other electronic device.
* suffers from claustrophobia or feels that he will be unable to lie still on his back in the PET camera.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12-08 (Actual); Primary Completion 2009-06-11 (Actual); Study Completion 2009-06-11 (Actual)

PRIMARY OUTCOMES:
Binding of PHNO, PET ligand, in each region of interest at each scan. | up to 48 hours
Percentage of PHNO, PET ligand, occupancy in each region of interest after a single oral dose of GSK618334 for each individual. | up to 48 hours
Time course of GSK618334 concentration in blood following a single oral dose. | up to 48 hours

SECONDARY OUTCOMES:
Adverse events and other safety assessments such as clinically relevant changes in electrocardiography (ECG); vital signs (blood pressure, heart rate); laboratory safety data and physical examination. | screening to follow-up
Measuring GSK618334 in the body (pharmacokinetic endpoints): PK parameters of GSK618334 Cmax, AUCinf, tmax. | up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 110269 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/110269?search=study&study_ids=110269#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 110269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register